CLINICAL TRIAL: NCT00657020
Title: Simultaneous fMRI/EEG of the 4 mg Nicotine Lozenge in Relief of Cognitive Impairment Associated With Nicotine Withdrawal
Brief Title: Functional Magnetic Resonance Imaging (fMRI) Investigation of Nicotine Withdrawal Symptoms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: S3250493
Record Dates: First submitted 2008-04-02; First posted 2008-04-14 (Estimated); Results first posted 2010-04-06 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2013-06

CONDITIONS: Smoking
Keywords: nicotine; therapy; fMRI/EEG; replacement
MeSH Terms: conditions — Smoking | interventions — Nicotine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nicotine lozenge (Experimental): Nicotine lozenge containing 4 mg of nicotine to be placed in mouth and suck to dissolution.
  Interventions: Drug: Nicotine
- Placebo lozenge (Placebo Comparator): Placebo lozenge to be placed in mouth and suck to dissolution.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nicotine — Nicotine lozenge containing 4 mg of nicotine
  Arms: Nicotine lozenge
Drug: Placebo — Placebo lozenge
  Arms: Placebo lozenge

SUMMARY:
A single center, double blind, randomized, placebo controlled, two-treatments, two-period crossover study conducted in adult smokers.

DETAILED DESCRIPTION:
The main objective of this study is to use blood oxygen level-dependent (BOLD) functional Magnetic Resonance Imaging (fMRI) in abstinent smokers to directly evaluate the effect of the 4 milligrams (mg) nicotine lozenge on brain activation associated with visual attention. The experimental task featured 3 conditions: 1. a highly demanding cognitive/attention task, 2. a simple cognitive/attention task, and 3. simply look at a '+' symbol. During the experiment these conditions are each presented a number of times in an alternating manner while acquiring images.

ELIGIBILITY:
Inclusion Criteria:

* Weight and size

  1. Body mass index (BMI) within the range 19.0-32.0 kg/m.
  2. Able to fit comfortably within the MR scanner.
* Smoking Status

  1. Cigarette smokers that consume their first manufactured cigarette (i.e., not self rolled cigarettes) within 30 min of waking.
  2. Individuals who have smoked regularly for at least a year.
* Females of childbearing potential who are, in the opinion of the investigator, practicing a reliable method of contraception.
* Understands and is willing, able and likely to comply with all study procedures and restrictions.
* Good general health with (in the opinion of the examining study doctor) no clinically significant and relevant abnormalities of medical history, physical examination or clinical laboratory test.
* Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.

Exclusion Criteria:

* Women who are pregnant or who have a positive urine pregnancy test or
* who are breast-feeding.
* Disease/Illness

  1. Any clinically significant medical history or abnormality found on physical examination, laboratory assessment or electrocardiogram (ECG) at screening which, in the opinion of the investigator, could interfere with the interpretation of efficacy or safety data or which otherwise would contraindicate participation in a clinical trial.
  2. Current or recent history or presence of a neurological diagnosis (not limited to but including for example, stroke, traumatic brain injury, carotid arterial sclerotic disease, epilepsy, space occupying lesions, multiple sclerosis, Parkinson's disease, vascular dementia, transient ischemic attack, schizophrenia, major depression etc.) that may influence the outcome or analysis of the scan results.
* Contraindications to MR scanning

  1. Intracranial aneurysm clips
  2. History of intra-orbital metal fragments that have not been removed by a doctor (as confirmed by orbital X-Ray).
  3. Inner ear implants.
  4. Tattoos with metal containing inks or piercings that can not be removed except those, which, in the opinion of the Investigator, will not interfere with the study procedures or compromise safety.
  5. History of claustrophobia or subject feels unable to lie still on their back for a period of 90 min in the MR scanner.
  6. Presence of a cardiac pacemaker or other electronic device or ferromagnetic metal foreign bodies in vulnerable positions as assessed by a standard pre-MRI questionnaire supported by plain X-Rays where appropriate.
* Prior/Concomitant Medication

  1. Use of any central nervous system (CNS) active, prescription medication within 14 days of first treatment visit.
  2. Use of any over the counter (OTC) medication within 14 days of each treatment visit except those, which, in the opinion of the Investigator, will not interfere with the study procedures or compromise safety. Paracetamol (up to 2 g) may be taken up to 24 hrs prior to each treatment visit.
  3. Current use of any nicotine replacement therapy.
* Clinical Study/Experimental Medication

  1. Participation in another clinical study or receipt of an investigational drug within 3 months of the first treatment visit.
  2. Previous participation in this study.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Substance abuse

  1. History of regular alcohol consumption exceeding an average weekly intake of more than 14 units per week for females, 21 units per week for males, or an average daily intake greater than 2 units for females and 3 units for males.
  2. Past history of drug abuse, excluding nicotine, or has tested positive for urine drugs of abuse at the screening or either treatment visit.
* Consumption of any alcoholic beverages within 24 hours of the treatment visits (as indicated by either a positive breath alcohol test or in the opinion of the Investigator).
* Consumption of large quantities of xanthine containing beverages (e.g., coffee, tea, cola, chocolate etc, more than an average of five cups or glasses per day).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2007-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 45 participants were screened, 22 were considered screen failures. Investigators identified brain regions showing significant blood oxygen-level dependent (BOLD) activation associated with attention in each participant using Functional Magnetic Resonance Imaging (fMRI). Hence, participants categorized into high/low attention conditions.
Groups:
- 4 mg Nicotine Lozenge Then Placebo Lozenge: Participants received nicotine lozenge containing 4 milligrams (mg) of nicotine in Period I and placebo lozenge in Period II.
- Placebo Lozenge Then 4 mg Nicotine Lozenge: Participants received placebo lozenge in Period I and nicotine 4 mg lozenge in Period II.
Period: PERIOD 1
Arm/Group | 4 mg Nicotine Lozenge Then Placebo Lozenge | Placebo Lozenge Then 4 mg Nicotine Lozenge
Started | 11 | 12
Completed | 11 | 11
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: PERIOD 2
Arm/Group | 4 mg Nicotine Lozenge Then Placebo Lozenge | Placebo Lozenge Then 4 mg Nicotine Lozenge
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Participants: All randomized participants who receive study treatments.
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.82 (8.428)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 18
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 23

OUTCOME MEASURES:

1. Primary Outcome: Percent Mean Change in Blood Oxygen-level Dependent (BOLD) Scores During Rapid Visual Information Processing (RVIP) Task
Description: In RVIP task, participant responded to consecutive sequences of three odd or three even numbers by pressing the corresponding response button as quickly and accurately as possible. During a control task, participant responded to single occurrences of the number "0". BOLD fMRI signals evaluated different brain regions of interest (ROI) during RVIP task. Brain ROIs identified were right and left anterior insula, anterior putamen, parietal cortex, premotor cortex, visual cortex, dorsal anterior cingulate cortex, substantia nigra and thalamus.
Time Frame: Approximately 2 hours post dose administration
Population: Number of participants with complete imaging data on both treatments (nicotine and placebo).
Measure: Mean (Standard Deviation); unit: Percentage change in BOLD signal
Groups:
- Nicotine Lozenge 1: Participants in low attention condition and received 4 mg of nicotine lozenge.
- Placebo Lozenge 1: Participants in low attention condition and received placebo lozenge.
- Nicotine Lozenge 2: Participants in high attention condition and received 4 mg of nicotine lozenge.
- Placebo Lozenge 2: Participants in high attention condition and received placebo lozenge.
Arm/Group | Nicotine Lozenge 1 | Placebo Lozenge 1 | Nicotine Lozenge 2 | Placebo Lozenge 2
Number analyzed (Participants) | 18 | 18 | 18 | 18
Percentage change in BOLD signal
  BOLD - Left Anterior Insula | 0.0 (0.21) | 0.2 (0.27) | 0.7 (0.48) | 0.7 (0.39)
  BOLD - Left Anterior Putamen | 0.0 (0.20) | 0.1 (0.36) | 0.3 (0.27) | 0.3 (0.34)
  BOLD - Left Dorsal Anterior Cingulate Cortex | 0.3 (0.39) | 0.4 (0.31) | 1.4 (0.70) | 1.0 (0.66)
  BOLD - Left Dorsolateral Pre-Frontal Cortex | 0.0 (0.29) | 0.1 (0.25) | 0.7 (0.77) | 0.7 (0.59)
  BOLD - Left Parietal Cortex | 0.3 (0.49) | 0.2 (0.37) | 1.5 (0.90) | 1.2 (0.59)
  BOLD - Left Premotor Cortex | 0.1 (0.27) | 0.1 (0.24) | 0.9 (0.69) | 0.7 (0.46)
  BOLD - Left Substantia Nigra/Ventral Tegemental | 0.1 (0.18) | 0.1 (0.29) | 0.4 (0.28) | 0.3 (0.33)
  BOLD - Left Thalamus | 0.1 (0.24) | 0.1 (0.36) | 0.5 (0.36) | 0.6 (0.39)
  BOLD - Left Visual Cortex | 0.9 (0.72) | 0.9 (0.73) | 1.6 (0.73) | 1.9 (0.87)
  BOLD - Right Anterior Insula | 0.0 (0.18) | 0.1 (0.24) | 0.5 (0.35) | 0.5 (0.40)
  BOLD - Right Dorsal Anterior Cingulate Cortex | 0.2 (0.34) | 0.2 (0.17) | 0.8 (0.57) | 0.8 (0.49)
  BOLD - Right Dorsolateral Pre-Frontal Cortex | 0.2 (0.45) | 0.2 (0.37) | 1.0 (0.85) | 0.8 (0.55)
  BOLD - Right Parietal Cortex | 0.2 (0.46) | 0.2 (0.52) | 1.1 (0.62) | 1.2 (0.72)
  BOLD - Right Premotor Cortex | 0.1 (0.47) | 0.2 (0.33) | 0.7 (0.61) | 0.8 (0.62)
  BOLD - Right Thalamus | -0.1 (0.22) | 0.0 (0.44) | 0.7 (0.44) | 0.6 (0.55)
  BOLD - Right Visual Cortex | 0.0 (0.44) | -0.1 (0.32) | 0.4 (0.43) | 0.3 (0.32)
Statistical Analysis 1: Comparison: Nicotine Lozenge 1 vs Placebo Lozenge 1; Region of Interest is left anterior insula; Test type: Superiority or Other; p = 0.2960, ANOVA
Statistical Analysis 2: Comparison: Nicotine Lozenge 2 vs Placebo Lozenge 2; Region of interest is left anterior insula; Test type: Superiority or Other; p = 0.3450, ANOVA
Statistical Analysis 3: Comparison: Nicotine Lozenge 1 vs Placebo Lozenge 1; Region of interest is left anterior putamen; Test type: Superiority or Other; p = 0.1192, ANOVA
Statistical Analysis 4: Comparison: Nicotine Lozenge 2 vs Placebo Lozenge 2; Region of interest is left anterior putamen; Test type: Superiority or Other; p = 0.6639, ANOVA
Statistical Analysis 5: Comparison: Nicotine Lozenge 1 vs Placebo Lozenge 1; Region of interest is left dorsal anterior cingulate cortex; Test type: Superiority or Other; p = 0.8295, ANOVA
Statistical Analysis 6: Comparison: Nicotine Lozenge 2 vs Placebo Lozenge 2; Region of interest is left dorsal anterior cingulate cortex; Test type: Superiority or Other; p = 0.0078, ANOVA
Statistical Analysis 7: Comparison: Nicotine Lozenge 1 vs Placebo Lozenge 1; Region of interest is left dorsolateral pre-frontal cortex; Test type: Superiority or Other; p = 0.7153, ANOVA
Statistical Analysis 8: Comparison: Nicotine Lozenge 2 vs Placebo Lozenge 2; Region of interest is left dorsolateral pre-frontal cortex; Test type: Superiority or Other; p = 0.8511, ANOVA
Statistical Analysis 9: Comparison: Nicotine Lozenge 1 vs Placebo Lozenge 1; Region of interest is left parietal cortex; Test type: Superiority or Other; p = 0.4228, ANOVA
Statistical Analysis 10: Comparison: Nicotine Lozenge 2 vs Placebo Lozenge 2; Region of interest is left parietal cortex; Test type: Superiority or Other; p = 0.0611, ANOVA
Statistical Analysis 11: Comparison: Nicotine Lozenge 1 vs Placebo Lozenge 1; Region of interest is left premotor cortex; Test type: Superiority or Other; p = 0.9879, ANOVA
Statistical Analysis 12: Comparison: Nicotine Lozenge 2 vs Placebo Lozenge 2; Region of interest is left premotor cortex; Test type: Superiority or Other; p = 0.2065, ANOVA
Statistical Analysis 13: Comparison: Nicotine Lozenge 2 vs Placebo Lozenge 2; Region of interest is left substantia nigra/ventral tegmental area; Test type: Superiority or Other; p = 0.1837, ANOVA
Statistical Analysis 14: Comparison: Nicotine Lozenge 1 vs Placebo Lozenge 1; Region of interest is left substantia nigra/ventral tegmental area; Test type: Superiority or Other; p = 0.8195, ANOVA
Statistical Analysis 15: Comparison: Nicotine Lozenge 1 vs Placebo Lozenge 1; Region of interest is left thalamus; Test type: Superiority or Other; p = 0.6420, ANOVA
Statistical Analysis 16: Comparison: Nicotine Lozenge 2 vs Placebo Lozenge 2; Region of interest is left thalamus; Test type: Superiority or Other; p = 0.7475, ANOVA
Statistical Analysis 17: Comparison: Nicotine Lozenge 1 vs Placebo Lozenge 1; Region of interest is left visual cortex; Test type: Superiority or Other; p = 0.9049, ANOVA
Statistical Analysis 18: Comparison: Nicotine Lozenge 2 vs Placebo Lozenge 2; Region of interest is left visual cortex; Test type: Superiority or Other; p = 0.1830, ANOVA
Statistical Analysis 19: Comparison: Nicotine Lozenge 1 vs Placebo Lozenge 1; Region of interest is right anterior insula; Test type: Superiority or Other; p = 0.5318, ANOVA
Statistical Analysis 20: Comparison: Nicotine Lozenge 2 vs Placebo Lozenge 2; Region of interest is right anterior insula; Test type: Superiority or Other; p = 0.9588, ANOVA
Statistical Analysis 21: Comparison: Nicotine Lozenge 1 vs Placebo Lozenge 1; Region of interest is right dorsal anterior cingulate cortex; Test type: Superiority or Other; p = 0.7551, ANOVA
Statistical Analysis 22: Comparison: Nicotine Lozenge 2 vs Placebo Lozenge 2; Region of interest is right dorsal anterior cingulate cortex; Test type: Superiority or Other; p = 0.7895, ANOVA
Statistical Analysis 23: Comparison: Nicotine Lozenge 1 vs Placebo Lozenge 1; Region of interest is right dorsolateral pre-frontal cortex; Test type: Superiority or Other; p = 0.9494, ANOVA
Statistical Analysis 24: Comparison: Nicotine Lozenge 2 vs Placebo Lozenge 2; Region of interest is right dorsolateral pre-frontal cortex; Test type: Superiority or Other; p = 0.4482, ANOVA
Statistical Analysis 25: Comparison: Nicotine Lozenge 1 vs Placebo Lozenge 1; Region of interest is right parietal cortex; Test type: Superiority or Other; p = 0.9343, ANOVA
Statistical Analysis 26: Comparison: Nicotine Lozenge 2 vs Placebo Lozenge 2; Region of interest is right parietal cortex; Test type: Superiority or Other; p = 0.7711, ANOVA
Statistical Analysis 27: Comparison: Nicotine Lozenge 1 vs Placebo Lozenge 1; Region of interest is right premotor cortex; Test type: Superiority or Other; p = 0.4755, ANOVA
Statistical Analysis 28: Comparison: Nicotine Lozenge 2 vs Placebo Lozenge 2; Region of interest is right premotor cortex; Test type: Superiority or Other; p = 0.3982, ANOVA
Statistical Analysis 29: Comparison: Nicotine Lozenge 1 vs Placebo Lozenge 1; Region of interest is right thalamus; Test type: Superiority or Other; p = 0.4622, ANOVA
Statistical Analysis 30: Comparison: Nicotine Lozenge 2 vs Placebo Lozenge 2; Region of interest is right thalamus; Test type: Superiority or Other; p = 0.4604, ANOVA
Statistical Analysis 31: Comparison: Nicotine Lozenge 1 vs Placebo Lozenge 1; Region of interest is right visual cortex; Test type: Superiority or Other; p = 0.2485, ANOVA
Statistical Analysis 32: Comparison: Nicotine Lozenge 2 vs Placebo Lozenge 2; Region of interest is right visual cortex; Test type: Superiority or Other; p = 0.1931, ANOVA

2. Secondary Outcome: Mean Response Time for Correct Responses During RVIP Task
Description: During the RVIP task, participants responded to consecutive sequences of three odd or three even numbers by pressing the corresponding response button as quickly and accurately as possible. During a control task, participants responded to single occurrences of the number "0". Mean response time for correct responses was determined.
Time Frame: Approximately 2 hours post dose administration
Population: Number of participants with complete imaging data on both treatments (nicotine and placebo).
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | Nicotine Lozenge 1 | Placebo Lozenge 1 | Nicotine Lozenge 2 | Placebo Lozenge 2
Number analyzed (Participants) | 22 | 22 | 22 | 22
milliseconds (msec) | 0.5 (0.05) | 0.5 (0.05) | 0.5 (0.08) | 0.5 (0.06)
Statistical Analysis 1: Comparison: Nicotine Lozenge 1 vs Placebo Lozenge 1; Null hypothesis considered the response time of treatments in comparison to be equal; Test type: Superiority or Other; p = 0.4535, ANOVA
Statistical Analysis 2: Comparison: Nicotine Lozenge 2 vs Placebo Lozenge 2; Null hypothesis considered the response time of treatments in comparison to be equal; Test type: Superiority or Other; p = 0.1811, ANOVA

3. Secondary Outcome: Mean Percentage of Correct Responses During RVIP Task
Description: Percentage of correct responses during RVIP task was determined
Time Frame: Approximately 2 hours post dose administration
Population: Number of participants with complete imaging data on both treatments (nicotine and placebo).
Measure: Mean (Standard Deviation); unit: Percentage of responses correct
Groups:
- Nicotine Lozenge 1: Participants in low attention conditions and received 4 mg of nicotine lozenge.
- Placebo Lozenge 1: Participants in low attention conditions and received placebo lozenge.
- Nicotine Lozenge 2: Participants in high attention conditions and received 4 mg of nicotine lozenge.
- Placebo Lozenge 2: Participants in high attention conditions and received placebo lozenge.
Arm/Group | Nicotine Lozenge 1 | Placebo Lozenge 1 | Nicotine Lozenge 2 | Placebo Lozenge 2
Number analyzed (Participants) | 22 | 22 | 22 | 22
Percentage of responses correct | 92.6 (5.27) | 91.1 (4.32) | 62.4 (18.51) | 54.1 (15.38)
Statistical Analysis 1: Comparison: Nicotine Lozenge 1 vs Placebo Lozenge 1; Null hypothesis considered treatments in comparison to be equal; Test type: Superiority or Other; p = 0.6261, ANOVA
Statistical Analysis 2: Comparison: Nicotine Lozenge 2 vs Placebo Lozenge 2; Null hypothesis considered treatments in comparison to be equal; Test type: Superiority or Other; p = 0.0106, ANOVA

4. Secondary Outcome: Percent Mean Change in BOLD Scores During Divided Attention (DIA) Task
Description: BOLD fMRI signals evaluated different brain ROIs during DIA task which comprised of three conditions: i) Sustained visual attention wherein participant responded to letter "s" every time it appeared in a continuous stream of letters on a screen; ii) Sustained auditory attention wherein participant responded to the number "8" each time in appeared in a continuous stream of numbers presented through headphones; iii) Divided attention task auditory and visual stimuli wherein participant responded to occurrences of "s" (visual) and "8" (auditory) simultaneously. Brain ROIs were right and left parietal cortex, visual cortex, superior occipital cortex and right premotor cortex.
Time Frame: Approximately 2 hours post dose admininstration
Population: Number of participants with complete imaging data on both treatments (nicotine and placebo).
Measure: Mean (Standard Deviation); unit: Percentage change in BOLD signal
Arm/Group | Nicotine Lozenge 1 | Placebo Lozenge 1 | Nicotine Lozenge 2 | Placebo Lozenge 2
Number analyzed (Participants) | 19 | 19 | 19 | 19
Percentage change in BOLD signal
  Left Parietal Cortex | 0.0 (0.39) | 0.1 (0.33) | 0.7 (0.44) | 0.6 (0.40)
  Left Superior Occipital Cortex | -0.1 (0.32) | 0.0 (0.28) | 0.4 (0.40) | 0.4 (0.33)
  Left Visual Cortex | -0.1 (0.48) | -0.1 (0.41) | 0.8 (0.42) | 0.6 (0.54)
  Right Parietal Cortex | -0.1 (0.55) | -0.1 (0.63) | 0.5 (0.45) | 0.5 (0.39)
  Right Premotor Cortex | 0.1 (0.35) | 0.2 (0.57) | 0.5 (0.33) | 0.7 (0.58)
  Right Superior Occipital Cortex | 0.0 (0.37) | 0.0 (0.46) | 0.5 (0.43) | 0.5 (0.53)
  Right Visual Cortex | 0.0 (0.54) | 0.0 (0.68) | 1.0 (1.13) | 1.2 (1.21)
Statistical Analysis 1: Comparison: Nicotine Lozenge 1 vs Placebo Lozenge 1; Region of interest is left parietal cortex; Test type: Superiority or Other; p = 0.5544, ANOVA
Statistical Analysis 2: Comparison: Nicotine Lozenge 2 vs Placebo Lozenge 2; Region of interest is left parietal cortex; Test type: Superiority or Other; p = 0.6716, ANOVA
Statistical Analysis 3: Comparison: Nicotine Lozenge 1 vs Placebo Lozenge 1; Region of interest is left superior occipital cortex; Test type: Superiority or Other; p = 0.7511, ANOVA
Statistical Analysis 4: Comparison: Nicotine Lozenge 2 vs Placebo Lozenge 2; Region of interest is left superior occipital cortex; Test type: Superiority or Other; p = 0.7959, ANOVA
Statistical Analysis 5: Comparison: Nicotine Lozenge 1 vs Placebo Lozenge 1; Region of interest is left visual cortex; Test type: Superiority or Other; p = 0.6418, ANOVA
Statistical Analysis 6: Comparison: Nicotine Lozenge 2 vs Placebo Lozenge 2; Region of interest is left visual cortex; Test type: Superiority or Other; p = 0.2205, ANOVA
Statistical Analysis 7: Comparison: Nicotine Lozenge 1 vs Placebo Lozenge 1; Region of interest is right parietal cortex; Test type: Superiority or Other; p = 0.5135, ANOVA
Statistical Analysis 8: Comparison: Nicotine Lozenge 2 vs Placebo Lozenge 2; Region of interest is right parietal cortex; Test type: Superiority or Other; p = 0.9781, ANOVA
Statistical Analysis 9: Comparison: Nicotine Lozenge 1 vs Placebo Lozenge 1; Region of interest is right premotor cortex; Test type: Superiority or Other; p = 0.3755, ANOVA
Statistical Analysis 10: Comparison: Nicotine Lozenge 2 vs Placebo Lozenge 2; Region of interest is right premotor cortex; Test type: Superiority or Other; p = 0.2612, ANOVA
Statistical Analysis 11: Comparison: Nicotine Lozenge 1 vs Placebo Lozenge 1; Region of interest is right superior occipital cortex; Test type: Superiority or Other; p = 0.8486, ANOVA
Statistical Analysis 12: Comparison: Nicotine Lozenge 2 vs Placebo Lozenge 2; Region of interest is right superior occipital cortex; Test type: Superiority or Other; p = 0.8318, ANOVA
Statistical Analysis 13: Comparison: Nicotine Lozenge 1 vs Placebo Lozenge 1; Region of interest is right visual cortex; Test type: Superiority or Other; p = 0.7554, ANOVA
Statistical Analysis 14: Comparison: Nicotine Lozenge 2 vs Placebo Lozenge 2; Region of interest is right visual cortex; Test type: Superiority or Other; p = 0.5421, ANOVA

5. Secondary Outcome: Mean Response Time for Correct Responses During DIA Task
Description: DIA task comprised of three conditions: i) Sustained visual attention wherein participant responded to letter "s" every time it appeared in a continuous stream of letters on a screen; ii) Sustained auditory attention wherein participant responded to the number "8" each time in appeared in a continuous stream of numbers presented through headphones; iii) Divided attention task auditory and visual stimuli wherein participant responded to occurrences of "s" (visual) and "8" (auditory) simultaneously. Mean response time for correct responses was determined.
Time Frame: Approximately 2 hours post dose administration
Population: Number of participants with complete imaging data on both treatments (nicotine and placebo).
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Nicotine Lozenge 1 | Placebo Lozenge 1 | Nicotine Lozenge 2 | Placebo Lozenge 2
Number analyzed (Participants) | 22 | 22 | 22 | 22
msec | 0.4 (0.04) | 0.5 (0.04) | 0.5 (0.04) | 0.5 (0.04)
Statistical Analysis 1: Comparison: Nicotine Lozenge 1 vs Placebo Lozenge 1; Null hypothesis considered response time of treatments in comparison to be equal; Test type: Superiority or Other; p = 0.1963, ANOVA
Statistical Analysis 2: Comparison: Nicotine Lozenge 2 vs Placebo Lozenge 2; Null hypothesis considered response time of treatments in comparison to be equal; Test type: Superiority or Other; p = 0.0959, ANOVA

6. Secondary Outcome: Mean Percentage of Correct Responses During DIA Task
Description: Mean percentage of correct responses during DIA task was determined.
Time Frame: Approximately 2 hours post dose administration
Population: Number of subjects with complete imaging data on both treatments (nicotine and placebo)
Measure: Mean (Standard Deviation); unit: Percentage of responses correct
Arm/Group | Nicotine Lozenge 1 | Placebo Lozenge 1 | Nicotine Lozenge 2 | Placebo Lozenge 2
Number analyzed (Participants) | 18 | 18 | 18 | 18
Percentage of responses correct | 48.2 (0.97) | 47.8 (1.15) | 96.9 (3.48) | 95.9 (3.61)
Statistical Analysis 1: Comparison: Nicotine Lozenge 1 vs Placebo Lozenge 1; Null hypothesis considered treatments in comparison to be equal; Test type: Superiority or Other; p = 0.5400, ANOVA
Statistical Analysis 2: Comparison: Nicotine Lozenge 2 vs Placebo Lozenge 2; Null hypothesis considered the treatments in comparison to be equal; Test type: Superiority or Other; p = 0.1800, ANOVA

ADVERSE EVENTS:
Time Frame: All adverse events encountered or spontaneously reported following administration of any investigational product (including washout product), or for up to 5 days after the last administration of investigational product were recorded.
Groups:
- Nicotine Lozenge: Participants in safety population received 4 mg of nicotine lozenge.
- Placebo Lozenge: Participants in safety population received placebo lozenge.
Arm/Group | Nicotine Lozenge | Placebo Lozenge
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 4/22 | 0/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine Lozenge (N=22) | Placebo Lozenge (N=23)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes